CLINICAL TRIAL: NCT04245306
Title: Pilot Evaluation of a New Computerized Test for Pragmatic Inferences in Children with Autism Spectrum Disorder Aged 8-12 Years Old
Brief Title: Pilot Evaluation of a New Computerized Test for Pragmatic Inferences in Children with ASD
Acronym: TIPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01721-56
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: pragmatic inferences; non-literal language; autism; attention-deficit; hyperactivity disorder; ADHD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Three groups of children are included to be compared, in order to test the primary and secondary hypothesis of this study :
  * A group of 25 children with autism spectrum disorders (ASD)
  * A larger group of 190 typically developing children (TD)
  * A group of 25 children with developmental language disorders (DLD)
  * A group of 25 children with attention-deficit/hyperactivity disorder (ADHD group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Children with Autism Spectrum Disorders (Experimental): A group of 25 children with autism spectrum disorders (ASD)
  Interventions: Other: computerized test for pragmatic inferences
- Typically Developing children (Active Comparator): A larger group of 150 typically developing children (TD)
  Interventions: Other: computerized test for pragmatic inferences
- Children with Developmental Language Disorders (Experimental): A group of 25 children with developmental language disorders (DLD)
  Interventions: Other: computerized test for pragmatic inferences
- children with attention-deficit/hyperactivity disorder (ADHD group) (Experimental): 25 children with attention-deficit/hyperactivity disorder (ADHD group)
  Interventions: Other: computerized test for pragmatic inferences

INTERVENTIONS:
Other: computerized test for pragmatic inferences — Computerized tests

SUMMARY:
This study aims to evaluate the relevance of a new computerized test for pragmatic inferences (TIPi) in children aged 8 to 12 YO, presenting a typical development, autism spectrum disorders, another neurodevelopmental condition and attention-deficit/hyperactivity disorder.

DETAILED DESCRIPTION:
By virtue of pragmatic inference-making, a listener can go above and beyond the linguistic meaning of the speaker's utterance in order to understand what the speaker intended to communicate. Such inferences allow the listener to understand inter alia irony, metaphor, indirect requests, scalar and ad-hoc implicatures. Autistic individuals have typically been described, by clinicians and language specialists, as tending towards having a literal understanding of language and as being deficient with respect to understanding a speaker's intended meaning, and these difficulties have a major impact on quality of life and social participation. Therefore, assessing these abilities seems essential, both for diagnosis purpose and to draw a clear description of an individual's functioning profile. Yet, no tool is available for children aged 8 to 12 in French. A new test named TIPi has been developed to resolve this issue. This new test is computerized and runs in a touch pad. The main goal of the present study is to evaluate the ability of the TIPi to discriminate autism spectrum disorders (ASD), attention-deficit/hyperactivity disorder (ADHD) children from typically developing (TD) children. Secondary goals are (i) to measure the typical development of these abilities in TD children in this age range, (ii) to assess the developmental link these skills might have with other cognitive of language abilities (mentalizing, cognitive flexibility, core language skills, central coherence), and (iii) to compare the pragmatic profile of ASD children with another neurodevelopmental condition: developmental language disorder, in order to test the relevance of this test for differential diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 8 and 12 years old
2. Native French speaker
3. Informed consent of the parents and children
4. [For ASD group] Diagnosis of ASD provided by a trained and entitled clinician
5. [For DLD group] Diagnosis of DLD provided by a trained and entitled clinician
6. [For ASD and DLD groups] IQ above 70
7. Intellectual efficiency within the norm (ITQ > 70), confirmed by objective results (psychometrics) in the participant's file, or collected if necessary within the framework of this study (using the WISC V);
8. Medical diagnosis of Attention Deficit Hyperactivity Disorder (ADHD) by a competent professional, confirmed by a parental assessment (ADHD-RS-IV)

Exclusion Criteria:

1. Uncorrected visual impairment
2. Uncorrected auditory impairment
3. Motor disability preventing the use of a touch pad
4. [For the TD group] Diagnosis of any neurodevelopmental or psychiatric condition
5. [For ASD group] Diagnosis of language disorder of attention disorder (ADHD)
6. [For DLD group] Diagnosis of ASD or ADHD
7. [For ADHD group] Diagnosis of ASD or DLD

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Discrimination power of the measure assessed by the dissociation of the developmental trajectories of children with ASD compared to TD children in the composite score of the TIPi. | One day
  The dissociation between the developmental trajectories of these two groups will be assessed by comparing the coefficients of the linear regressions linking performance in the TIPi (composite score) and chronological age in these two groups.

SECONDARY OUTCOMES:
Sensitivity of the TIPi composite score (measuring pragmatic inferencing) to typical development in the targeted age range: 8 to 12 years oldin the targeted age range: 8 to 12 years old | One day
  Sensitivity to age of the TIPi composite score is assessed by the alpha coefficient of the regression analysis linking the composite score to chronological age in the TD group.
The TIPi composite score provides additional information compared to other cognitive assessments typically provided in the global assessment of children with ASD | One day
  The predictive power of the best fitted multiple regression model explaining this measure by - jointly - performances in language task, mentalizing task, cognitive flexibility task, central coherence task and age (this predictive power being measured by the adjusted R2 of the model).
Discrimination power of the measure assessed by the dissociation of the developmental trajectories of children with ASD compared to children with DLD in the composite score of the TIPi. | One day
  The dissociation between the developmental trajectories of these two groups will be assessed by comparing the coefficients of the linear regressions linking performance in the TIPi (composite score) and chronological age in these two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No